CLINICAL TRIAL: NCT06716957
Title: Effectiveness of Schroth Exercises and Dynamic Stabilization Exercises in Individuals With Adolescent Idiopathic Scoliosis: a Randomized Controlled Trial.
Brief Title: The Effectiveness of Different Exercises in Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar18
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Scoliosis; Adolescent Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): Schroth exercises
  Interventions: Other: Schroth exercise
- exercise (Experimental): Schroth exercise and dynamic stabilization exercises
  Interventions: Other: Schroth exercise; Other: Dynamic Stabilization exercises

INTERVENTIONS:
Other: Schroth exercise — Exercises will be given in lying, sitting and standing positions. In each exercise, elongation of the spine will be ensured and the person will be positioned according to the type of scoliosis. Exercises will be given progressively in supine, prone, side sitting, sitting and standing positions. In each exercise, elongation of the spine will be ensured and the person will be positioned according to the upper and lower extremities. Progress in the exercises will be made positionally by increasing the number of repetitions and the number of rotational breathing during the exercise.
Other: Dynamic Stabilization exercises — The dynamic neuromuscular stabilization group will receive developmental postures based on developmental kinesiology. It will involve a supine 3month Position, side-lying Position, Quadruped, oblique sitting, bear position, squat Position. Each position will be performed for 30-60 s for five reps, active exercise 5-10 reps under supervision for two days/week, and unsupervised for 3 days/week for 12 weeks
  Arms: exercise

SUMMARY:
The aim of this study is to examine the effectiveness of stabilization exercises integrated with Schroth exercises on quality of life, trunk rotation angle, body awareness and sleep quality in young people with scoliosis.

DETAILED DESCRIPTION:
The study will include adolescents who come to Bursa Eforfiz Healthy Living Center for outpatient treatment. Participants will be selected from adolescents between the ages of 10-17. Participants will first read the voluntary consent form and if they agree to participate in the study, they will then be evaluated by a physiotherapist. First, the demographic information of the participants will be questioned and then the evaluation will be done in a single session. Participants will be randomly divided into two groups. These will be the control group and the exercise group. Both groups will perform the determined exercises for 8 weeks in a private clinic with a physiotherapist. Only scales, forms and surveys with Turkish reliability and validity studies will be used in the evaluation methods. The surveys will be uploaded to the digital environment and filled in with the physiotherapist according to the participant's answers. All collected data will be scored by the physiotherapist in accordance with the scoring systems and the obtained data will be evaluated using the SPSS program.

ELIGIBILITY:
Inclusion Criteria:

* Being between 9-17 years of age
* Having a primary curve between 10-40 degrees according to the Cobb method
* Having typical S or C scoliosis
* Being willing to participate in the study
* Having the cognitive capacity to cooperate with the guidance of a physiotherapist

Exclusion Criteria:

* Having a BMI over 30 kg/m2
* Having any neurological, orthopedic, cardiopulmonary disorders other than the diagnosis of scoliosis
* Having had any injuries related to the musculoskeletal system in the last 6 months
* Being unable to fulfill exercise requirements for any reason

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Scoliosis Research Society-22 | 14 weeks
  It is a scoliosis-specific, valid and reliable quality of life scale that questions pain, body image perception, function/activity, mental health, and satisfaction with treatment. A minimum of 1 point (worst) and a maximum of 5 points (best) are taken for each question. Scoring is obtained by dividing the total score from each section by the number of questions in that section. As a result of the scoring, it is accepted that the higher the score, the higher the quality of life.
Walter Reed Visual Assessment | 14 weeks
  It is a valid scale consisting of 7 questions, each of which includes 5 visuals and evaluates the physical deformity perceived by the patients.The selected images are scored as the lowest "1" and the highest "5", and the highest total score is 35 and the lowest is 5. It is accepted that the higher the score, the more negative-evil perception of the deformity.
Pittsburgh Sleep Quality Index | 14 weeks
  The scale includes a total of 24 questions. 19 of these questions are self-evaluation questions, and 5 of them are answered by the individual's spouse or a roommate. These 5 questions are used for clinical information only and are not included in the scoring. The scale questions that determine sleep quality include various factors related to sleep quality. These questions are to determine sleep duration, sleep latency, and the frequency and severity of specific sleep-related problems; 18 items were grouped as 7 component scores. The total score ranges from 0 to 21. A high total score indicates poor sleep quality. The scale does not indicate the presence of sleep disorders or the prevalence of sleep disorders. However, it is stated that a total score of 5 and above indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Sude Asya ALŞAN MOVAHHEDİ, Study Chair — Uskudar University
Locations (1):
- Bursa Eforfiz Healthy Living Center, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almahmoud OH, Baniodeh B, Musleh R, Asmar S, Zyada M, Qattousah H. Overview of adolescent idiopathic scoliosis and associated factors: a scoping review. Int J Adolesc Med Health. 2023 Nov 21;35(6):437-441. doi: 10.1515/ijamh-2023-0166. eCollection 2023 Dec 1. PMID 37982659
- [Background] Mohamed N, Acharya V, Schreiber S, Parent EC, Westover L. Effect of adding Schroth physiotherapeutic scoliosis specific exercises to standard care in adolescents with idiopathic scoliosis on posture assessed using surface topography: A secondary analysis of a Randomized Controlled Trial (RCT). PLoS One. 2024 Apr 30;19(4):e0302577. doi: 10.1371/journal.pone.0302577. eCollection 2024. PMID 38687741
- [Background] Gan X, Liu X, Cai D, Zhang R, Li F, Fang H, Huang J, Qiu C, Zhan H. Wearable accelerometers reveal objective assessment of walking symmetry and regularity in idiopathic scoliosis patients. PeerJ. 2024 Jul 16;12:e17739. doi: 10.7717/peerj.17739. eCollection 2024. PMID 39035168